CLINICAL TRIAL: NCT00284674
Title: Prospective Clinical Evaluation of Three Prosthesis Re-cap, M2a-Magnum and C2a-taper.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Frederiksberg University Hospital (Other)
Responsible Party: Principal Investigator, Arne Borgwardt, MD, Frederiksberg University Hospital
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: KF-01-287.591
Record Dates: First submitted 2006-01-31; First posted 2006-02-01 (Estimated); Last update posted 2017-03-24 (Actual); Status verified 2017-03

CONDITIONS: Patients Undergoing a THR
MeSH Terms: interventions — Hip Prosthesis

INTERVENTIONS:
Device: Hip prosthesis (re-cap, m2a-magnum and C2a-taper)

SUMMARY:
This evaluation is being conducted to evaluate the performance of thee prosthesis.

ELIGIBILITY:
Inclusion Criteria:

* Good general health of age (ASA I-II)
* DEXA-scanning: lower limit for a 55 years old man
* MRI normal vitality in caput
* Willing to return for follow-up evaluations
* Exclusion Criteria:
* Subjects displaying any of the following contra-indications shall be excluded from this evaluation:
* Inability to co-operate with and complete the study
* Collum < 2 cm
* Large cysts in caput
* Mismatch between caput acetabulum
* Caput necrosis

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2006-03 (Actual); Primary Completion 2007-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Arne Borgwardt, M.D., Study Director — Frederiksberg University Hospital
Locations (1):
- Frederiksberg University Hospital, Copenhagen, Frederiksberg, Denmark

REFERENCES:
- [Derived] Borgwardt A, Borgwardt L, Zerahn B, Daugaard H, Borgwardt L, Ribel-Madsen S. A Randomized Seven-Year Study on Performance of the Stemmed Metal M2a-Magnum and Ceramic C2a-Taper, and the Resurfacing ReCap Hip Implants. J Arthroplasty. 2018 May;33(5):1412-1420. doi: 10.1016/j.arth.2017.11.061. Epub 2017 Dec 5. PMID 29276121